CLINICAL TRIAL: NCT01779414
Title: STAT-ED: Suicidal Teens Accessing Treatment After an Emergency Department Visit
Acronym: STAT-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CINC-2012-3660
Record Dates: First submitted 2013-01-02; First posted 2013-01-30 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Suicide
Keywords: Suicide Ideation
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (No Intervention): Participants in this arm of the study will receive a standard, usual care psychological risk assessment by a social worker and then recommended to a mental health referral.
- STAT-ED Intervention (Experimental): Participants in this group will receive a motivational interview conducted by a study trained social worker, where the social worker and the family will discuss the participants issues, thoughts and feelings about receiving treatment, barriers to treatment and methods of overcoming those barriers. The study trained social worker will also make a referral for a mental health follow-up for the patient.
  Interventions: Other: STAT-ED Intervention

INTERVENTIONS:
Other: STAT-ED Intervention — Participants in this group will receive a motivational interview conducted by a study trained social worker, where the social worker and the family will discuss the participants issues, thoughts and feelings about receiving treatment, barriers to treatment and methods of overcoming those barriers. The study trained social worker will also make a referral for a mental health follow-up for the patient.
  Arms: STAT-ED Intervention

SUMMARY:
This study looks to implement a novel intervention (STAT-ED) for children who screen positive to suicide ideation. The intervention looks to collect data from several different measures and then randomize participants into one of two groups: a control group where the participant will be set up with a mental health referral from a psychiatric social worker; or if randomized into the STAT-ED intervention, the adolescent and parent will receive a brief motivational interview, barrier reduction discussion, referral and limited case management by the study social worker to enhance outpatient mental health follow up after discharge from the ED.

The hypothesis of the study is patients who are randomized into the STAT-ED intervention group will have a significantly higher rate of initiating mental health treatment and will attend more mental health treatment sessions in the two months after the ED visit compared with adolescents in the control group. Secondary aims of this study look to determine whether the effectiveness of the STAT-ED intervention differs by age, gender, or ethnicity; and evaluate predictors and mediators of mental health treatment engagement.

DETAILED DESCRIPTION:
The STAT-ED study is a two site study conducted by Cincinnati Children's Hospital and Nationwide Children's Hospital that is looking to test the effectiveness of a brief treatment engagement intervention termed Suicidal Teens Accessing Treatment After an ED Visit (STAT-ED) for adolescents seeking treatment in the ED for non-psychiatric concerns but identified via systematic screening as being at risk for suicide. In this study, investigators from both institutions will recruit and randomize 160 adolescents (80 per site) to either(a) the STAT-ED intervention or (b) enhanced usual care group (EUC). The EUC group consist of a brief consultation by an ED social worker and a mental health referral for the participant facilitated by the Psychiatric Intake Response Center. The STAT-ED intervention targets family engagement, problem solving, motivational interviewing, assistance with referral and limited case management during the transition from the ED to outpatient care with the goal of maximizing the initiation of mental health treatment and aftercare among youth screening positive for previously unrecognized suicide risk. A study trained research coordinator who is blinded to the participants treatment allocation will contact the participants via telephone at two months and six months post ED visit in order to ascertain initiation and attendance of the mental health follow-up, as well as an assessment of suicidal ideation and depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who arrive in the ED who are between the ages of 12-17 years old
* Screen positive on the Ask Suicide-Screening Questions (ASQ) tool
* Have had no contact with a mental health provider in the 90 days preceding the current ED visit
* Are stable as determined by vital signs and triage criteria (triage levels 2-5)

Exclusion Criteria:

* Patients who present in the ED with a chief complaint of suicidal behavior will be excluded to comply with the requirements of the RFA.
* Those who present in the ED with a primary or secondary psychiatric concern
* Those without access to a telephone/cell phone
* Those unable to adequately understand the study process
* Those families unable to speak or read English adequately to participate in study procedures
* Patients who have altered mental status either due to illness or medication (pain medications)
* Patients who live greater than 100 miles away form the enrolling site

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
STAT-ED Intervention Superior to EUC Group | Three years
  Adolescents receiving the STAT-ED intervention will have a significantly higher rate of initiating mental health treatment and will attend more mental health treatment sessions in the two months after the ED visit compared with adolescents in the EUC condition. STAT-ED will also be superior to the EUC arm in reducing suicidal ideation and depression symptoms at two months and six months.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Grupp-Phelan, M.D., M.P.H., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Grupp-Phelan J, Stevens J, Boyd S, Cohen DM, Ammerman RT, Liddy-Hicks S, Heck K, Marcus SC, Stone L, Campo JV, Bridge JA. Effect of a Motivational Interviewing-Based Intervention on Initiation of Mental Health Treatment and Mental Health After an Emergency Department Visit Among Suicidal Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1917941. doi: 10.1001/jamanetworkopen.2019.17941. PMID 31860104